CLINICAL TRIAL: NCT03193164
Title: Effects of Physical Therapy With Neuromuscular Electrical Stimulation in Patients With Septic Shock: a Randomised Crossover Clinical Trial Protocol.
Brief Title: Neuromuscular Electrical Stimulation and Septic Shock
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: This study had to be suspended due to COVID-19 Pandemic.
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ada Clarice Gastaldi, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: USP 2017-1
Record Dates: First submitted 2017-06-05; First posted 2017-06-20 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Shock, Septic
Keywords: Electric Stimulation Therapy; Endothelial Progenitor Cells.
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Intervention Model Description: This study will be randomized crossover clinical trial.
Who Masked: Investigator
Masking Description: The blood samples will be mask analyses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): Neuromuscular Electrical Stimulation (NMES) and after decubitus position with the limbs raised without NMES.
  Interventions: Device: Neuromuscular Electrical Stimulation; Other: Decubitus Position with the limbs raised to 20º
- group 2 (Sham Comparator): Decubitus Position with the limbs raised to 20º without NMES and after NMES.
  Interventions: Device: Neuromuscular Electrical Stimulation; Other: Decubitus Position with the limbs raised to 20º

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — The patient will be positioned on a headboard at 30° in the decubitus position with the limbs raised to 20°. The location of the electrical current will be cleared with trichotomy when necessary. Adhesive electrodes 90 x 50 mm will be positioned in the gastrocnemius. The stimulator device will be the Neurodyn II (Ibramed, Sao Paulo, Brazil) to provide symmetrical biphasic pulses of 50 Hz, 250 µsec pulse duration, 2 seconds on (1 second of time of rise and 1 second of time of decay), and 5 seconds of rest during 30 minutes at an intensity capable of generating visible contractions and articular motion.
  Other Names: Functional Electrical Stimulation
Other: Decubitus Position with the limbs raised to 20º — The patient position will be the same used for intervention protocol (headboard to 30°, decubitus position with the limbs raised to 20°) for 30 minutes, without NMES.

SUMMARY:
The study will investigate the effects of neuromuscular electrical stimulation (NMES) in patients with septic shock. The objective of this study will be investigate the effects of neuromuscular electrical stimulation (NMES) in patients with septic shock.

DETAILED DESCRIPTION:
The study will investigate the effects of neuromuscular electrical stimulation (NMES) in patients with septic shock.

It will be a randomised crossover clinical trial. Thirty-one patients will enrolled.The study will be divided in two phases, the first will be held in the first 72 hours of septic shock and the second after three days of first assessment. Patients will be selected, randomly, to the intervention Protocol (NMES) and control (positioning). After this procedure the patients will be allocated in Group 1 (NMES and control) or group 2 (control and NMES), with a wash-out period of 4 to 6 hours in between .

The main outcome will be the study of mobilization of endothelial progenitor cells (EPCs). The secondary outcome will be the metabolic and hemodynamic data. Linear mixed model will be used for analysis of dependent variables and estimated values of the mean of the differences of each effect.

The results of this study will allow better understanding of the effects of NMES in patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:The patients admitted to the intensive care unit will be considered eligible if:

* they present in the first 72 hours the diagnosis of septic shock according to the international consensus definition of septic shock, and
* stable hemodynamics through fluid resuscitation, and
* vasoactive drugs and mechanical ventilation.

Exclusion Criteria:The exclusion criteria will be patients aged less than 18 years and greater than 65 years, pregnant women, brain death, neuromuscular diseases, use of pre-existing neuromuscular blocker in the last 24 hours, prior to the study protocol.

* Contraindications for the use of NMES: fractures, burns and skin lesions, systemic vascular impairment diseases such as systemic lupus erythematosus, thromboembolic disease, deep vein thrombosis (which was not therapeutically anticoagulated for a time greater than 36 hours), lower limb amputations, cardiac pacemaker, thrombocytopenia less than 20,000/mm3, BMI greater than 35 kg/m2, important lower extremity oedema, agitation and/or signs of pain during the electrical stimulation.
* Contraindications to begin or continue NMES procedure: Mean arterial blood pressure less than 65 mmHg, use of vasopressor >50% of the maximum dose (dopamine >12.5 µg/kg per minute; vasopressin >0.02U/min and norepinephrine >1 µg/kg per minute), heart rate <50 or >140 bpm, arrhythmias with hemodynamic consequences, myocardial ischemia, temperature <34 or >39oC, intracranial pressure >20 cmH2O, decrease in 10% of SpO2 baseline value or <88% for more than one minute.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2021-01-29 (Estimated)

PRIMARY OUTCOMES:
Change of counts of Endothelial Progenitor Cells (EPCs) | It will be taken at the baseline and at the end of the each intervention.The data will be collected in two phases, the first will be held in the first 72 hours of septic shock and the second after three days of first assessment.
  Change of counts of mobilization of endothelial progenitor cells will be quantified by cytometry markers:+/CD133+/CD45-, CD34+/CD133+/CD45-/VEDFR2 e CD45-/VEGFR2+.

SECONDARY OUTCOMES:
Change of Oxygen consumption (VO2), Carbon dioxide production (VCO2) and Resting energy expenditure (REE). | It will be taken at the baseline and at the end of the each intervention.The data will be collected in two phases, the first will be held in the first 72 hours of septic shock and the second after three days of first assessment.
  Indirect calorimetry is a noninvasive method that analyzes the amount of heat generated. by the whole body according to the substrate utilization. The data provided by calorimetry are: Resting Energy Expenditure (REE) which is calculated from the amount of oxygen consumed (VO2) and carbon dioxide produced (VCO2) through the respiratory gases.

OTHER OUTCOMES:
Change of hemodynamic and respiratory variables | It will be taken at the baseline and at the end of the each intervention.The data will be collected in two phases, the first will be held in the first 72 hours of septic shock and the second after three days of first assessment.
  It will be measured heart rate, blood pressure, oxygen saturation and breathing frequency.
Change of Cirtometry | Patients will be measured at the first, the third and the seventh day
  Measurements of the circumference of the gastrocnemius muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Ada C Gastaldi, PhD, Principal Investigator — Ribeirão Preto Medicine School - University of São Paulo
Locations (1):
- Hospital das Clínicas, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available immediately following publication and for five years.
Access Criteria: The data will be available from the principal investigator upon reasonable request.

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Stefanou C, Karatzanos E, Mitsiou G, Psarra K, Angelopoulos E, Dimopoulos S, Gerovasili V, Boviatsis E, Routsi C, Nanas S. Neuromuscular electrical stimulation acutely mobilizes endothelial progenitor cells in critically ill patients with sepsis. Ann Intensive Care. 2016 Dec;6(1):21. doi: 10.1186/s13613-016-0123-y. Epub 2016 Mar 11. PMID 26969168
- [Background] Duda DG, Cohen KS, Scadden DT, Jain RK. A protocol for phenotypic detection and enumeration of circulating endothelial cells and circulating progenitor cells in human blood. Nat Protoc. 2007;2(4):805-10. doi: 10.1038/nprot.2007.111. PMID 17446880
- [Background] Fadini GP, Losordo D, Dimmeler S. Critical reevaluation of endothelial progenitor cell phenotypes for therapeutic and diagnostic use. Circ Res. 2012 Feb 17;110(4):624-37. doi: 10.1161/CIRCRESAHA.111.243386. PMID 22343557
- [Derived] Lago AF, Basile-Filho A, de Oliveira AS, de Souza HCD, Dos Santos DO, Gastaldi AC. Effects of physical therapy with neuromuscular electrical stimulation in acute and late septic shock patients: A randomised crossover clinical trial. PLoS One. 2022 Feb 17;17(2):e0264068. doi: 10.1371/journal.pone.0264068. eCollection 2022. PMID 35176099